CLINICAL TRIAL: NCT04224558
Title: Autologous Hematopoietic Stem Cell Transplantation for Refractory Crohn's Disease
Brief Title: Stem Cell Transplantation in Crohn's Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Ziring, Associate Director, Pediatric IBD Center, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00051458
Record Dates: First submitted 2018-04-04; First posted 2020-01-13 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Mesna; Cyclophosphamide; Filgrastim; Leukapheresis; fludarabine; fludarabine phosphate; Methylprednisolone; Methylprednisolone Hemisuccinate; Diphenhydramine; Acetaminophen; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HSCT after mobilization and conditioning (Experimental): Mobilization and leukopheresis allow for stem cell harvest. Then conditioning is provided prior to stem cell transplantation, followed by post-transplant conditioning.
  Interventions include:
  1. Stem cell mobilization
  2. Leukopheresis
  3. Preparative regimen
  4. Peripheral blood stem cell infusion
  5. Post-PBSC infusion conditioning
  Interventions: Drug: Mesna; Drug: Cyclophosphamide; Drug: Filgrastim; Procedure: Apheresis catheter placement; Procedure: Leukapheresis; Drug: Fludarabine; Drug: Methylprednisolone; Drug: Diphenhydramine; Drug: Acetaminophen; Drug: anti-thymocyte globulin (rabbit); Drug: lymphocyte immune globulin; Biological: Peripheral Blood Stem Cell Infusion; Drug: Cytoxan

INTERVENTIONS:
Drug: Mesna — Stem Cell Mobilization: Infused according to institutional guidelines;
  Post-PBSC Infusion Conditioning: Mesna provided with Cytoxan according to institutional protocol.
  Other Names: Mesnex
Drug: Cyclophosphamide — Stem Cell Mobilization:
  Cyclophosphamide (CY) infused intravenously over 1 hour: 50 mg/kg (25 mg/kg/day on 2 consecutive days)
  Other Names: Cytoxan; Neosar
Drug: Filgrastim — Stem Cell Mobilization: Filgrastim (G-CSF) 10 mcg/kg SC will start 5 days after the last dose of CY and will end the day before the last leukapheresis;
  Post-PBSC Infusion Conditioning: Filgrastim administered intravenously 5 mcg/kg IV starting day + 5, continue until ANC of >1000/μL
  Other Names: Neupogen; Granix
Procedure: Apheresis catheter placement — Subjects will require placement of an Apheresis catheter by Intervention Radiologists on the day of collection of stem cells.
Procedure: Leukapheresis — Leukapheresis will be performed on a continuous flow separator machine according to institutional guidelines to target 3-8 x 10^6 CD34+ cells/kg body weight.
Drug: Fludarabine — Preparative/Conditioning Regime Fludarabine given as 30 mg/m2 per dose x 4 days, beginning on day -6.
  Other Names: Fludara
Drug: Methylprednisolone — Preparative/Conditioning Regime r-ATG pre-medication according to institutional guidelines
  Other Names: solu-medrol
Drug: Diphenhydramine — Preparative/Conditioning Regime r-ATG premedication according to institutional guidelines
  Other Names: Benadryl
Drug: Acetaminophen — Preparative/Conditioning Regime r-ATG premedication according to institutional guidlines
  Other Names: Tylenol
Drug: anti-thymocyte globulin (rabbit) — Preparative/Conditioning Regime r-ATG administered intravenously: 2.5 mg/kg/dose IV over 6 hours on specified days (day -6,-4,-2); ); total 3 doses=7.5 mg/kg.
  Other Names: thymoglobulin
Drug: lymphocyte immune globulin — Preparative/Conditioning Regime In patients who develop severe allergic reactions to rATG (Thymoglobulin), it may be substituted by horse ATG (hATG, ATGAM, Pharmacia & Upjohn, Kalamazoo, MI). The recommended dose of hATG is 25 mg/kg/day for 3 doses.
  Other Names: ATGAM
Biological: Peripheral Blood Stem Cell Infusion — PBSC (peripheral blood stem cell) infusion on day 0 as per institutional guidelines.
Drug: Cytoxan — Post-PBSC Infusion Conditioning Cytoxan infused intravenously: 50mg/kg/day x 2 days. Infused over 2 hours with adequate hydration or according to institutional guidelines.
  Other Names: Cyclophosphamide

SUMMARY:
Unfortunately, some patients with Crohn's disease (CD) fail to respond to the best clinical treatments and some only experience temporary benefit. For severe Crohn's disease, there is an experimental treatment called "high dose immunoablation" followed by autologous hematopoietic stem cell transplantation (HSCT). This study removes over active lymphocytes (immunoablation) and replaces them using blood stem cells that have been taken from the patient's own body. The aim of the study is to reset or reprogram the patient's immune system to its state prior to diagnosis.

DETAILED DESCRIPTION:
The treatment of Crohn's disease has proven to be quite efficacious in the majority of patients with the timely use of combination therapies for remission induction (corticosteroids and/or biologics) and maintenance of disease control (immunosuppressives and/or biologics). However, a proportion of patients fail to achieve complete and long term disease control and often require multiple intestinal surgeries with a risk of developing short bowel syndrome. Lymphoablation followed by hematopoietic stem cell transplantation to rescue the immune system has been proposed as an alternative strategy to induce long term disease control in this high-risk population. It has been demonstrated that despite the potential toxicity and morbidity associated with the procedure, the benefit-risk ratio is favorable. Hence, the investigators propose to offer HSCT to selected CD patients and to study mechanisms of reducing T cell autoreactivity which will hopefully lead to more focused therapeutic approaches in the future.

This is an open-label, non-randomized, non-blinded, prospective study in therapeutic refractory Crohn's patients, failing conventional therapy.

The primary objective is to evaluate the safety and potential clinical benefit of lymphoablation followed by autologous HSCT rescue in therapy refractory CD. Death (transplant-related mortality, TRM) and severe toxicity (≥ grade 3 toxicity; NCI Toxicity Criteria version 4.0) within the first 6 months after HSCT will be monitored to meet this end-point.

SECONDARY OBJECTIVES

1. To evaluate the incidence of HSCT related complications, i.e. viral reactivations (CMV, Adenovirus, EBV, BK virus) or fungal infections.
2. To evaluate the impact of HSCT on quality of life and school productivity.
3. To elucidate the underlying mechanism involved in the observed benefit of HSCT on CD.

First, the safety will be evaluated by the amount of related adverse events. All adverse events will be recorded in a standardized way and their relationship to the study protocol will be assessed at various short and long term time points.

Second, to determine clinical benefit, the percentage of patients in sustained disease remission at 0, 2, 4, 6, 12 and 24 months post HSCT will be determined. Sustained disease remission is defined as a Crohn's Disease Activity Index (CDAI) < 150 without the use of corticosteroids. In addition, mucosal healing will be assessed during ileocolonoscopy at 6 and 12 months following HSCT using the CD endoscopic index (SES).

SECONDARY ENDPOINTS

- Change in Crohn's disease endoscopic index after 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 13-28 years are eligible
2. Confirmed diagnosis of active Crohn's disease:

   1. Diagnosis of Crohn's disease based on typical radiological appearances and / or typical histology at least 6 months prior to screening.
   2. Active disease at the time of registration to the trial, defined as

   i) PCDAI > 30, and ii) Two of the following:
   1. elevated CRP
   2. endoscopic evidence of active disease confirmed by histology
   3. clear evidence of active small bowel Crohn's disease on CT or MR enterography.
3. Unsatisfactory course despite 3 immunosuppressive agents (usually azathioprine, methotrexate and infliximab, adalimumab and/or certolizumab) in addition to corticosteroids. Patients should have relapsing disease (i.e. 1 exacerbation/year) despite thiopurines, methotrexate and/or infliximab/adalimumab/certolizumab maintenance therapy or clear demonstration of intolerance / toxicity to these drugs.
4. Current problems unsuitable for surgery or patient at risk for developing short bowel syndrome.
5. Accepted by a majority of the members of the combined IBD Center as an appropriate candidate (see Selection description below).
6. Informed consent

   1. Prepared to undergo additional study procedures as per trial schedule
   2. Patient has undergone intensive counseling about risks

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during the study, in women of childbearing age. Unwillingness of using appropriate contraceptive measures in males.
2. Concomitant severe disease

   1. renal: creatinine clearance < 30 mL/min (measured or estimated)
   2. cardiac: clinical evidence of refractory congestive heart failure; left ventricular ejection fraction < 40% by cardiac echo; chronic atrial fibrillation necessitating oral anticoagulation; uncontrolled ventricular arrhythmia; pericardial effusion with hemodynamic consequences as evaluated by an experienced echo cardiographer
   3. pulmonary: diffusion capacity <40%
   4. psychiatric disorders including active drug or alcohol abuse
   5. concurrent or recent history of malignant disease (excluding non-melanoma skin cancer)
   6. uncontrolled hypertension, defined as resting systolic blood pressure ≥ 140 and/or resting diastolic pressure ≥ 90 despite at least 2 anti-hypertensive agents.
   7. any infection with HIV, HTLV-1 or 2, hepatitis viruses, or any other infection the investigators consider a contraindication to participation.
   8. other chronic disease causing significant organ failure.
3. Infection or risk thereof:

   1. Current clinical relevant abscess or significant active infection.
   2. Perianal fistula without free drainage. Perianal fistulas is not an exclusion provided there is natural free drainage or a seton suture(s) have been placed.
   3. History of tuberculosis or at current increased risk of tuberculosis
   4. Quantiferon Gold test result or other investigations that the investigators regard as evidence of active tuberculosis.
   5. Abnormal chest X-ray (CXR) consistent with active infection or neoplasm.

6) Significant malnutrition: Body Mass Index (BMI) ≤ 18, serum albumin < 20 g/l.

7) Previous poor compliance. 8) Concurrent enrollment in any other protocol using an investigational drug or hematopoietic growth factor up to four weeks before study entry.

Ages: 13 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mucosal healing | Change from pre-HSCT (baseline) to 6 months and 12 months post HSCT
  Change mucosal healing as determined by the simple endoscopic score for crohn's disease (SES-CD). The SES-CD assesses the size of mucosal ulcers, the ulcerated surface, the endoscopic extension and the presence of stenosis. Each are measured on a scale of 0-3 and are summed to create a total score. For total score, 0-2 indicates remission, 3-6 indicates mild endoscopic activity, 7-15 indicates moderate endoscopic activity, and > 15 indicates severe endoscopic activity.
Change in erythrocyte sedimentation rate (SED rate) | Change from pre-HSCT (baseline) to 2, 4, 6, 12, and 24 months post HSCT
  Change in SED rate (mm/hour)
Change in fecal calprotectin concentration | Change from pre-HSCT (baseline) to 2, 4, 6, 12, and 24 months post HSCT
  Change in fecal calprotectin concentration
Change in C reactive protein (CRP) | Change from pre-HSCT (baseline) to 2, 4, 6, 12, and 24 months post HSCT
  Change in C reactive protein (CRP)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 months post HSCT
  Number of treatment-emergent adverse events (including death (transplant related mortality, TRM) and severe toxicity (≥ grade 3 toxicity; NCI Toxicity Criteria version 4.0)
Incidence of HSCT Related Complications | Up to 24 months post HSCT
  The incidence of HSCT related complications, i.e. viral reactivations (CMV, Adenovirus, EBV, BK virus) or fungal infections.
Change in clinical measures of sustained remission | Up to 24 months post HSCT
  Change in CDAI score (Crohn's Disease Activity Index). The CDAI measure the signs, symptoms, and history of Crohn's Disease based on the past 7 days. The index measures abdominal pain, stools per day, general wellbeing, HCT, ESR, Albumin, height, weight, abdominal exam, perirectal disease, and extra-intestinal manifestations each scaled between 0-10. The sum of these measures creates a total score between 0-100 with the higher score representative of more disease activity.

SECONDARY OUTCOMES:
Change in quality of life | 0, 2, 4, 6, 12 and 24 months post HSCT
  Change in score on the IMPACT-III Questionnaire (A Quality of Life Questionnaire for Children with Inflammatory Bowel Disease) after HSCT. It is a self-report measure with 35 closed questions encompassing six proposed domains: Bowel Symptoms (7 items), Systemic Symptoms (3 items), Social Functioning (12 items), Body Image (3 items), Treatment/Interventions (3 items), and Emotional Functioning (7 items). The IMPACT-III uses 5-point Likert scale ranging from 1 to 5 for all answers. The outcome score ranges from 35 to 175, with higher scores suggesting better quality of life.
Change in school and work productivity | 0, 2, 4, 6, 12 and 24 months post HSCT
  Change in school productivity and activity impairment as determined by the modified Work Productivity and Activity Impairment (WPAI) Index score. The Modified WPAI yield four types of scores: absenteeism (school time missed), presenteeism (impairement at school), school productivity (overall work impairment/absenteeism plus presenteeism), and activity impairement. WPAI outcomes are expressed as impairement percentages, with higher numbers indicating greater impairement and less productivity.
Change in thymopoiesis after HSCT | 0, 2, 4, 6, 12 and 24 months post HSCT
  the amount of T-cell receptor excision circles (TREC) will be determined. TRECs are excision circles of DNA excised during the process of T cell receptor (TCR) rearrangement. Since these TRECs do not replicate during cell division, they can also be a measure for recent thymic emigrants.
Change in T-cell repertoire after HSCT using spectratyping | 0, 2, 4, 6, 12 and 24 months post HSCT
  The CDR3 (complement determining region) of the TCRβ chain is the most variable region of the TCR and is generated by recombination of the variable, diversity and joining region of the DNA. The length of this region differs between different T-cell clones due to nucleotide transferases or removed nucleotides during recombination, and the variability of these lengths can be used to estimate thymic diversity. This variability can be determined by electrophoresis, after amplification of this region by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: David Ziring, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No